CLINICAL TRIAL: NCT02162342
Title: Quantification of Kinematics and Muscle Activity Patterns of the Upper Extremities of Individuals With Motor Disabilities
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Isabella Shvartz, MD, Hadassah Medical Organization
Other Study IDs: Upper_Extremety- HMO-CTIL
Record Dates: First submitted 2014-06-11; First posted 2014-06-12 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Diagnosis and Follow up on Upper Extremity Interventions
Keywords: upper extremity; muscle activity; kinematics; motion capture; Electromyography
MeSH Terms: conditions — Disease | interventions — Braces

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (1):
- Rehabilitative intervention: Surgical intervention, orthotics or injections of muscle/nerve medications as prescribed by the treating physician and unrelated to the study.
  Interventions: Other: Rehabilitative treatment

INTERVENTIONS:
Other: Rehabilitative treatment — Surgical intervention, orthotics or injections of muscle/nerve medications as prescribed by the treating physician and unrelated to the study.
  Other Names: Corrective surgery; orthotics; injections of muscle/nerve medications

SUMMARY:
The subjet is sitting on a chair and in front of him an adjustable (height) table with a glass of water. 17 passive reflective markers are placed on his upper extremities and torso. The subject is requested to reach the glass (once with the right hand and then with the left hand) and bring it to the mouth and drink. Then the subject put the glass back at the starting position. This is performed twice for each hand. In the second part, the same trial is repeated but muscle activity is recorded with surface electromyography.

ELIGIBILITY:
Inclusion Criteria:

* motor impairment following stroke, multiple sclerosis, cerebral palsy, traumatic brain injury, spina bifida, poliomyelitis, neuropathy
* Able to understand and sign an informed consent form independently.

Exclusion Criteria:

* Unable to hold or lift a glass
* pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: stroke, multiple sclerosis, cerebral palsy, traumatic brain injury, spina bifida, poliomyelitis, neuropathy
Sampling Method: Probability Sample
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
joint angle | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel